CLINICAL TRIAL: NCT06712654
Title: A Phase 2b, Randomized, Double-Blinded, Placebo-Controlled, Multicenter Study to Evaluate the Safety, Tolerability, and Serum Phosphate Lowering Effect of Fixed Dosed AP306 in Patients Receiving Maintenance Hemodialysis with Hyperphosphatemia
Brief Title: A Study to Evaluate Safety, Tolerability and Efficacy of AP306 At Fixed Doses in Patients with Hyperphosphatemia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alebund Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AP306-HP-02
Record Dates: First submitted 2024-11-27; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Hyperphosphatemia; Chronic Kidney Disease Requiring Hemodialysis
MeSH Terms: conditions — Hyperphosphatemia | interventions — BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- AP306 (Experimental): A blood phosphate-lowering medication with a novel mechanism
  Interventions: Drug: AP306 75mg TID; Drug: AP306 100mg TID; Drug: AP306 125mg TID; Drug: AP306 125mg BID; Drug: AP306 150mg BID
- Placebo of AP306 (Placebo Comparator)
  Interventions: Drug: Placebo TID

INTERVENTIONS:
Drug: AP306 75mg TID — receiving orally AP306 75mg (one tablet), three times a day
  Arms: AP306
Drug: AP306 100mg TID — receiving orally AP306 100 mg (one tablet), three times a day.
  Arms: AP306
Drug: AP306 125mg TID — receiving orally AP306 125 mg (one tablet), three times a day
  Arms: AP306
Drug: AP306 125mg BID — receiving orally AP306 125 mg (one tablet), three times a day, among which one is a placebo tablet
  Arms: AP306
Drug: AP306 150mg BID — receiving orally AP306 150 mg (one tablet), three times a day, among which one is a placebo tablet
  Arms: AP306
Drug: Placebo TID — receiving orally one placebo tablet of AP306, three times a day
  Arms: Placebo of AP306

SUMMARY:
The goal of this clinical trial is to learn if AP306 could work in the patients receiving maintenance hemodialysis with elevated blood phosphate. The main questions it aims to answer are:

* Does AP306 lower blood phosphate levels when the participants take a fixed dose of AP306?
* What medical problems do the participants have when taking AP306?

The researchers will compare AP306 to a placebo (a look-alike substance that contains no drug) to see if AP306 works to treat hyperphosphatemia.

The participants will:

* Stop all using blood phosphate-lowering drugs, and
* Take AP306 or a placebo three times a day for 12 weeks.

If the participant has a blood phosphate level above a certain level, they will receive additional treatment to lower the blood phosphate level.

ELIGIBILITY:
Important Inclusion Criteria:

1. Who signes a written informed consent form (ICF) and is willing to comply with all study requirements in the study
2. Who is receiving a stable hemodialysis regimen, which is defined as a frequency of three times per week for at least 12 weeks before the ICF sign off, and doesn't plan to change in the study
3. Who has a dialysis adequacy, assessed by single pooled Kt/V (SpKt/V, estimated with blood urea) ≥1.20, at screening
4. If the participant is receiving any of the following therapies, their doses are stable for at least 4 weeks before the ICF sign off visit: phosphate-lowering products other than phosphate binders, active vitamin D and analogs or nutritional vitamin D, calcimimetics, calcitonin, and P-glycoprotein inhibitors or inducers
5. Who has a blood phosphate level within the study-required range

Important Exclusion Criteria:

1. Pregnant or breastfeeding
2. Scheduled for a living donor kidney transplant in the next 6 months, planned change to peritoneal dialysis or home hemodialysis in the study; planned relocation to another dialysis center in the study
3. Any history of a non-pharmacological parathyroid intervention within 6 months prior to the ICF sign off, or planned parathyroid intervention in the study
4. Uncontrolled blood calcium abnormality
5. Uncontrolled blood intact parathyroid hormone abnormality
6. Hemoglobin <9 mg/dL (90 g/L)
7. Acute hepatitis or significant chronic liver disease
8. Any clinically significant GI disorders within 4 weeks prior to the ICF sign off; or any history of gastrectomy; or any GI tract surgery, excluding appendectomy and polypectomy, within 12 weeks prior to the ICF sign off
9. Uncontrolled hypertension
10. Hospitalization for cardiac or cardiocerebrovascular disease within 24 weeks prior to the ICF sign off
11. Significant abnormalities of QT interval and heart rhythm on an electrocardiograph (ECG) test
12. Any active infection or infestation or any treatment with antibiotics within 2 weeks prior to the ICF sign off
13. History or presence of malignancy within 3 years prior to the ICF sign off, except basal cell skin cancer, in-situ carcinoma of the cervix, and in-situ prostate cancer
14. Concomitant use of moderate or strong cytochrome P450 (CYP) 3A inhibitors or inducers within 2 weeks or 5 half-lives, whichever is longer, prior to the ICF sign off (topical use is allowed)
15. Treatment with any investigational medication or medical device within 30 days prior to the ICF sign off

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-04-10 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of AP306 assessed by serum phosphate lowering | 12 weeks
  The change in serum phosphate from the baseline to the end of treatment or before the initiation of rescue therapy

OTHER OUTCOMES:
To evaluate the overall safety of AP306 assessed by incidence of treatment-emergent adverse events | 15 weeks
  All adverse events occurred after the study treatment initiation will be collected and their nature, frequency, and severity will be assessed.

IPD SHARING:
Plan to Share IPD: Undecided
The study will enroll part of participants from China. Sharing of individual participant data from them is not possible due to the Personal Information Protection Law of the People's Republic of China (Presidential Decree No. 91, August 2021). The IPD sharing will be decided later.